CLINICAL TRIAL: NCT01917448
Title: Low-dose Spinal Morphine for Post-Thoracotomy Pain After Video-Assisted Thoracoscopic Surgery: A Prospective Randomized Double-Blind Controlled Trial
Brief Title: Low-dose Spinal Morphine for Post-Thoracotomy Pain After Video-Assisted Thoracoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2556
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Video-assisted Thoracoscopic Surgery
Keywords: postoperative pain; spinal morphine; video-assisted thoracoscopic surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): The skin will be injected with local anesthetic without spinal block
  Interventions: Other: control
- Spinal morphine (Active Comparator): 0.15 mg spinal morphine
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — spinal morphine 0.15 mg
  Arms: Spinal morphine
Other: control — Patient receive only local infiltration without spinal analgesia
  Arms: Control

SUMMARY:
One-thirds of patients underwent video-assisted thorascopic surgery still have severe pain. Therefore we want to demonstrate weather 0.15 mg spinal morphine would reduce 24 hour postoperative requirement comparing to control group.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologist) physical status I to III,
* Undergoing elective video-assisted thoracoscopic surgery at Siriraj and Thammasart Hospitals
* capable of using a patient-controlled analgesia (PCA) machine
* understanding the numeric rating scale (NRS) score for pain assessment.

Exclusion Criteria:

* history of allergy to the study drugs
* bleeding disorder
* infection of the back
* refusing spinal anesthesia
* history of cerebrovascular disease
* using postoperative ventilator support were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Total post-operative morphine requirement. | 48 hours

SECONDARY OUTCOMES:
Pain after surgery | 48 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided